CLINICAL TRIAL: NCT02557217
Title: A Phase II Randomised, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety and Tolerability of Oral NP202 in Adults Who Have Left Ventricular Systolic Dysfunction Following Myocardial Infarction
Brief Title: NP202 for Treatment of Post -STEMI Left Ventricular Systolic Dysfunction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armaron Bio Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP202-002; ACTRN12615000609550 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2015-09-07; First posted 2015-09-23 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NP202 (Experimental): 1000mg oral NP202 daily for 90 days
  Interventions: Drug: NP202
- Placebo (Placebo Comparator): Oral placebo daily for 90 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NP202 — Active
  Arms: NP202
Other: Placebo — Placebo
  Other Names: Microcellulose
  Arms: Placebo

SUMMARY:
NP202 is an experimental drug being developed by Armaron Bio Pty Ltd for potential use as a treatment for people after they have had a heart attack (MI).

DETAILED DESCRIPTION:
After someone has a MI, their heart 'remodels', which means that it changes in size and shape. This damage can lead to it being weaker and less efficient, and ultimately to major heart problems. There are some drugs currently available which help prevent remodelling and are used for treatment post-MI. However, there is still a high rate of remodelling and major heart problems in people post-MI. NP202 works in a different way to the drugs that are currently approved, and has been shown in animal studies to prevent post-MI remodelling.

This study will assess NP202 versus placebo on remodelling over a 3 month treatment period, with 1 month follow up

ELIGIBILITY:
Inclusion Criteria:

* Have had a confirmed ST elevation myocardial infarction (STEMI) in the previous 5 days, which met all of the following criteria;

  * ≥ 0.2mV ST elevation in 2 or more V1 - V6 leads with presentation in a maximum of 12 hours of onset of symptoms
  * Troponin levels >10 x upper limit of normal (ULN) at the site's local laboratory.
  * Successful revascularisation by Percutaneous Coronary Intervention (PCI)
* Have left ventricular dysfunction post STEMI as evidenced by left ventricular ejection fraction (LVEF) ≤40% confirmed by echocardiogram at screening.
* Are receiving guideline-directed medical therapy for acute MI and post-MI left ventricular (LV) dysfunction according to national cardiology society/heart association STEMI guidelines.

Exclusion Criteria:

* Known cardiomyopathy or heart failure prior to MI.
* Cardiogenic shock and/or systolic blood pressure <85mmHg at Screening.
* Clinical history of ejection fraction ≤40% prior to this MI, or multiple prior MIs.
* Daily use of non-steroidal anti-inflammatory drugs (NSAIDs) and/or cyclooxygenase-2 (COX-2) inhibitors in the past month.
* Presence of device/hardware incompatible with MRI
* Estimated glomerular filtration rate (eGFR) <30ml/min
* Liver function tests 3 x ULN due to non-cardiac disease
* Have received any investigational research agent within 30 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by Change from baseline in left ventricular end systolic volume index (LVESVi) | From baseline to 3 months post MI
  Change from baseline in left ventricular end systolic volume index (LVESVi) as assessed by MRI at 3 months

SECONDARY OUTCOMES:
Efficacy as measured by Change from baseline in LV end diastolic volume index (LVEDVi) | From baseline to 3 months post MI
  Change from baseline in LV end diastolic volume index (LVEDVi) as assessed by MRI at 3 months.
Efficacy as measured by Change from baseline in LV ejection fraction (LVEF) | From baseline to 3 months post MI
  Change from baseline in LVEF as assessed by MRI at 3 months.
Efficacy as measured by Change from baseline in LV diastolic function | From baseline to 3 months post MI
  Changes from baseline in LV diastolic function based on LV peak filling rate as assessed by MRI at 3 months.
Efficacy as measured by Change from baseline in relative infarct size | From baseline to 3 months post MI
  Change from baseline in relative infarct size as a percent of LV mass as assessed by late contrast enhancement MRI at 3 months.

OTHER OUTCOMES:
Safety as assessed by occurrence of adverse events (AE) | From baseline to end of study (4 months)
  All AE occurring during the study will be recorded
Safety as assessed by changes in laboratory results | At Baseline, Week 2, and Months 1, 2, 3 and 4
  Biochemistry, haematology, prostate specific antigen (PSA), urinalysis
Safety as assessed by changes in physical examination | At Baseline, Week 2, and Months 1, 2, 3 and 4
  Changes in physical examination finding including vital signs (heart rate, blood pressure, respiratory rate, temperature)
Safety as assessed by changes in 12-lead electrocardiograms (ECGs). | At Baseline, Week 2, and Months 1, 2, 3 and 4
  Changes in ECG intervals
Trough levels of NP202 in plasma | At Baseline, Week 2 and at Months 1, 2 and 3
  Concentrations of NP202 in plasma in a subset of 30 subjects.
Efficacy as assessed by laboratory biomarkers | At Baseline and Months 1, 2 and 3
  Absolute values and changes from baseline in serum biomarker levels (Troponin I, Troponin T, high sensitivity C reactive protein (hs-CRP) and N-terminal of the prohormone brain natriuretic peptide (NT-proBNP)

CONTACTS AND LOCATIONS:
Overall Officials: Grant McLachlan, Study Director — Sponsor GmbH
Locations (1):
- John Hunter Hospital, Newcastle, New South Wales, Australia

REFERENCES:
- [Derived] Boyle AJ, Schultz C, Selvanayagam JB, Moir S, Kovacs R, Dib N, Zlotnick D, Al-Omary M, Sugito S, Selvarajah A, Collins N, McLachlan G. Calcium/Calmodulin-Dependent Protein Kinase II Delta Inhibition and Ventricular Remodeling After Myocardial Infarction: A Randomized Clinical Trial. JAMA Cardiol. 2021 Jul 1;6(7):762-768. doi: 10.1001/jamacardio.2021.0676. PMID 33851966